CLINICAL TRIAL: NCT02114463
Title: Comparison of Two Kinds of Postoperative Analgesia After Amputation:a Randomized Clinical Trial
Brief Title: Comparison of Two Kinds of Postoperative Analgesia After Amputation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, bo xu, associate chief physician, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Phantom limb pain
Record Dates: First submitted 2014-04-08; First posted 2014-04-15 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-03

CONDITIONS: Pain; Complications
Keywords: Local analgesia system; Ropivacaine; Analgesic efficacy after operation; Postoperative
MeSH Terms: conditions — Pain | interventions — Ropivacaine; Flurbiprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Local analgesic (Experimental): This group uses local analgesia infusion pump of 0.2% ropivacaine 360ml through periarticular infiltration for postoperative analgesia.
  Interventions: Procedure: Local analgesic; Drug: ropivacaine
- Intravenous analgesic (Active Comparator): This group is treated with intravenous electronic analgesia pump infusion of flurbiprofen axetil 250mg,palonosetron 0.5mg,pentazocine 240mg.dezocine 30mg.
  Interventions: Procedure: Intravenous analgesic; Drug: flurbiprofen

INTERVENTIONS:
Procedure: Local analgesic — Patient will be performed under combined lumbar plexus and sciatic nerve block with 0.33% ropivacaine.At the end of surgery,two catheters are left in the wound.One is intraarticular and the other is on the surface of articular cavity.And then a pump elastomeric infusion pump will be connected with the catheters, which runs 5mL every hours.
  Arms: Local analgesic
Procedure: Intravenous analgesic — People in this group will also receive an anesthesia of combined lumbar plexus and sciatic nerve block with 0.33% ropivacaine.An intravenous electronic analgesia pump infusion of flurbiprofen axetil 250mg,palonosetron 0.5mg,pentazocine 240mg.dezocine 30mg will will provide postoperative pain management.The patients will received a 2 mL/h continuous basal infusion and 1 mL boluses with a lockout time of 30 min after a 5 mL Loading dose at the end of the surgery.
  Arms: Intravenous analgesic
Drug: ropivacaine — 0.2% ropivacaine
  Arms: Local analgesic
Drug: flurbiprofen — flurbiprofen axetil 250mg,palonosetron 0.5mg,pentazocine 240mg.dezocine 30mg
  Arms: Intravenous analgesic

SUMMARY:
Pain after amputation is a significant problem among amputees. Phantom limb pain may appear in up to 85% of patients and is usually resistant to a wide variety of treatments.It is believed that regional anesthesia, by preventing the establishment of central sensitization, may play a role in reducing the incidence of acute and chronic pain. Therefore the investigators will compare two methods of postoperative analgesic after after amputation by their efficiency and complication.

DETAILED DESCRIPTION:
Peripheral nerve transection results in an afferent nociceptive barrage that initiates spinal cord hyperexcitability with expansion of the receptive fields of dorsal horn neurons that respond to the nearest intact afferents. These neuroplastic changes are believed to be responsible for the development of postsurgical chronic pain syndromes, including phantom limb and stump pain.At present, there are no randomized studies with sample sizes that ensure power, or blinded for end-point assessment,to support the evidence on pharmacological and non-pharmacological treatments of Pain after amputation. Consequently, our study was designed to arrive at clear conclusions about treatment efficacy and to give stronger recommendations for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of American Association of anesthetists（ASA）Grade 1 or 2
2. Aged between 18 and 65 years
3. Undergoing elective total knee replacement

Exclusion Criteria:

1. Mental illness can not match
2. Nerve block, epidural anesthesia contraindicated
3. People who have Slow-type arrhythmias
4. History of chronic headaches and long-term use of analgesic drugs
5. People who were postoperative consciousness, language or hearing impaired

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
pain | 72 hours postoperation
  Up to 72 hours after operation,postoperative pain visual analogue scale(VAS) scores are used to evaluate the level of pain.

SECONDARY OUTCOMES:
Phantom pain | three months postoperation
  Investigators asked the patient wether there is phantom pain at three months after surgery
complication | 72 hours postoperation
  Investigators document the incidence of nausea,vomiting,headache,urinary retention and et al

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Military Region General Hospital, Department of Anesthesiology, Guangzhou, Guangdong, China